CLINICAL TRIAL: NCT05743764
Title: A Multicenter, Randomized, Double Blind, Restasis®-Controlled Non-inferiority, Moisview® Eye Drops Controlled Superiority, Phase III Study to Evaluate the Efficacy and Safety of HU007 Eye Drops in Patients with Dry Eye Syndrome
Brief Title: HU007 in Patients with Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HUC2-007_P3-2
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HU007 (Experimental): Cyclosporine 0.02%, trehalose 3%
  1 drop b.i.d at 12hr interval for 12 weeks
  Interventions: Drug: HU007
- Restasis (Active Comparator): Cyclosporine 0.05%
  1 drop b.i.d at 12hr interval for 12 weeks
  Interventions: Drug: Restasis
- Moisview (Active Comparator): trehalose 3%
  1 drop b.i.d at 12hr interval for 12 weeks
  Interventions: Drug: Moisview Eye drop

INTERVENTIONS:
Drug: HU007 — cyclosporine 0.02%, trehalose 3%
  Arms: HU007
Drug: Restasis — cyclosporine 0.05%
  Arms: Restasis
Drug: Moisview Eye drop — trehalose 3%
  Arms: Moisview

SUMMARY:
A multicenter, Randomized, Double blind, Restasis®-controlled Non-inferiority, Moisview® Eye Drops Controlled Superiority, Phase III Study to Evaluate the Efficacy and Safety of HU007 Eye Drops in Patients with Dry Eye Syndrome

ELIGIBILITY:
Inclusion Criteria

* Age over 19
* Corneal staining score(Oxford grading) ≥ 2 and Schirmer test ≤ 10mm/5min (If Schirmer test = 0mm/5min, Nasal stimulation schirmer test ≥ 3mm/5min) and TBUT test ≤10 in at least one of both eyes
* Patients who have had more than one symptom of dry eye disease for at least 3 month before screening visit
* Best corrected visual acuity of 0.2 or higher in both eyes
* Those who voluntarily decided to participate and agreed in writing to comply with the precautions

Exclusion Criteria:

* Patients with clinically significant ocular disorders affected the test result
* Current or recent patients used dry eye syndrome medications (topical or systemic) that may affect the status
* SBP ≥140mmHg or DBP ≥ 90mmHg or HbA1c > 9%
* Wearing contact lenses within 72 hr prior to screening visit or during clinical trial
* Pregnancy or Breastfeeding
* Patient with a history of glaucoma, or intraocular pressure of 25mmHg or higher at least one eyes
* Patient with autoimmune disease (e.g. sjogren's syndrome)
* Patients with a history of corneal transplant or neurotrophic keratitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in corneal staining score | 12weeks
  Change in corneal staining score assessed on Oxford grading at 12 weeks compared to baseline
  - Oxford grading: 0(Absent) to 5(Severe)

SECONDARY OUTCOMES:
Change from baseline in corneal staining score | 4, 8weeks
  Change in corneal staining score assessed on Oxford grading at 4, 8 weeks compared to baseline
Change from baseline in conjuctival staining score | 4, 8, 12weeks
  Change in conjuctival staining score assessed on Oxford grading at 4, 8, 12 weeks compared to baseline
Change from baseline in strip meniscometry score | 4, 8, 12weeks
  Change in strip meniscometry score at 4, 8, 12 weeks compared to baseline
Change from baseline in TBUT score | 4, 8, 12weeks
  Change in TBUT score at 4, 8, 12 weeks compared to baseline
Change from baseline in SPEED dry eye questionnaire score | 4, 8, 12weeks
  Change in SPEED dry eye questionnaire score at 4, 8, 12 weeks compared to baseline
Time to achieve 100% clearance in corneal staining | 12weeks
  Time to achieve 100% clearance in corneal staining up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun young Hyun, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Gyeongsang National University Hospital, Jinju, South Korea

IPD SHARING:
Plan to Share IPD: No